CLINICAL TRIAL: NCT03894124
Title: Pharmacokinetics of Plasma Doravirine Once Daily Over 72 Hours Following Drug Intake Cessation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Imperial College London (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRF001; 2019-000978-33 (EudraCT Number)
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — doravirine

STUDY DESIGN:
Intervention Model Description: Single cohort pharmacokinetic (PK) study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study intervention (Other): Pifeltro® (doravirine 100mg) daily dose for 7 days
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — Non-nucleoside reverse transcriptase inhibitor. Administered as film coated tablet.
  Other Names: Pifeltro

SUMMARY:
Study to assess the pharmacokinetics of plasma doravirine once daily over 72 hours following drug intake cessation at steady-state in healthy volunteers

DETAILED DESCRIPTION:
The administration of combination antiretroviral therapy (cART) to HIV-infected patients has been associated with a dramatic reduction in AIDS-related morbidity and mortality. The key to successful HIV drug treatment is adhering to the prescribed combination every day. The approval of single tablet combinations (STRs) provides HIV care providers with a "one tablet once a day" therapy, making adherence much easier for patients. However, in HIV therapy, successful adherence also means attention to intervals between doses or dietary restrictions. Ideally, to guarantee long-term virological response, HIV-infected patients should take their cART every day at the same time. However, cART is for life and doses can be forgotten or delayed. For this study 14 healthy volunteers will receive Pifeltro® (doravirine 100mg tablets) daily for 7 days to reach steady state. Following the last dose samples will be taken for pharmacokinetic testing over 72 hours.

The incidence of adverse events between enrolment to the study (day 1) and last visit (day 20-23) will be recorded.

Blood, urine and faecal samples from study subjects will be taken for use in planned exploratory research and for use in future research:

Analyses looking at genes which affect drug disposition (pharmacogenomics); the impact of doravirine intake on platelet function and markers of platelet and endothelial cell activation; metabolic changes associated with doravirine.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females.
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive
5. ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
6. Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 4 weeks after the study. Any contraception method must be used consistently, in accordance with the approved product label and for at least 4 weeks after discontinuation of IMP.
7. Men who have partners who are women of childbearing potential must be using an adequate method of contraception to avoid pregnancy in their partner throughout the study and for a period of at least 4 weeks after the study. Any contraception method must be used consistently, in accordance with the approved product label and for at least four weeks after discontinuation of IMP.
8. Willing to consent to their personal details being entered onto the TOPS database
9. Willing to provide proof of identity by photographic ID at screen and any subsequent visit
10. Registered with a GP in the UK

Exclusion Criteria:

1. Any clinically significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B surface antigen or C antibody
4. Positive blood screen for HIV-1 or 2 by antibody/antigen assay
5. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
6. History or presence of allergy to the study drugs and their components
7. Current or recent (within three months) gastrointestinal disease
8. Known intolerance of lactose monohydrate, sunset yellow aluminium lake (E110), and patients with galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
9. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
10. Exposure to any investigational drug (or placebo) or participation in a clinical study involving the donation of blood samples within three months of first dose of study drug
11. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
12. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least four weeks after the end of the treatment period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliot ER, Cerrone M, Challenger E, Else L, Amara A, Bisdomini E, Khoo S, Owen A, Boffito M. Pharmacokinetics of dolutegravir with and without darunavir/cobicistat in healthy volunteers. J Antimicrob Chemother. 2019 Jan 1;74(1):149-156. doi: 10.1093/jac/dky384. PMID 30272231
- [Background] Wilby KJ, Eissa NA. Clinical Pharmacokinetics and Drug Interactions of Doravirine. Eur J Drug Metab Pharmacokinet. 2018 Dec;43(6):637-644. doi: 10.1007/s13318-018-0497-3. PMID 30047107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Intervention
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Fourteen (14) participants completed are considered sufficient to allow for relevant conclusions to be drawn, given experience from similar studies conducted previously.
Arm/Group | Study Intervention
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 33 [22 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 14
Median BMI [Median (Full Range); unit: kg/m2] | 23.3 [19.8 to 34.3]

OUTCOME MEASURES:

1. Primary Outcome: Steady State Plasma Concentrations of Doravirine After Drug Intake Cessation up to 72 Hours Post-dose.
Description: Following cessation of daily doravirine, plasma concentrations of drug to be taken before last dose and at 11 further timepoints over 72 hours. Blood samples were collected pre-dose and at 2, 4, 8, 12, 24, 30, 36, 48, 60 and 72 h post-dose
Time Frame: 72 hours from treatment cessation; days 7-10 inclusive from enrolment
Population: Plasma concentrations of doravirine after drug intake cessation up to 72 hours post-dose were investigated in population of participants for the study
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Study Intervention
Number analyzed (Participants) | 14
ng*hr/mL
  Doravirine steady-state PK parameters measured over 24h AUC 0-24h | 18354 [16395 to 21410]
  Doravirine steady-state PK parameters measured over 24h AUC 0-72h | 26338 [23080 to 31743]

2. Primary Outcome: Steady State Plasma Concentrations of Doravirine After Drug Intake Cessation up to 72h Post-dose
Description: Following cessation of daily dorovirine, plasma concentrations of drug to be taken before last dose and at 11 further timepoints over 72 hours. Blood samples were collected at pre-dose and at 2,4,8,12,24,30,36,47,60 and 72h post-dose
Time Frame: 72 hours from treatment cessation; days 7-10 inclusive from enrolment
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Study Intervention
Number analyzed (Participants) | 14
ng*hr/mL
  Cmax 0-24h | 1286 [1162 to 1488]
  Cmax 0-72h | 1286 [1188 to 1462]

3. Primary Outcome: Steady State Plasm Concentrations of Doravirine After Drug Intake Cessation up to 72 Hours Post-dose
Description: Following cessation of daily dorovirine, plasma concentrations of drug to be taken before last dose and at 11 further timepoints over 72 hours. Blood samples were collected pre-dose and at 2, 4, 8, 12, 24, 30, 36, 48, 60 and 72h post-dose
Time Frame: 72 hours from treatment cessation; days 7-10 inclusive from enrolment
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Study Intervention
Number analyzed (Participants) | 14
ng*hr/mL
  Ctrough at 24 h | 420 [373 to 526]
  Ctrough at 72 h | 39 [33 to 61]

4. Primary Outcome: Steady State Plasma Concentrations of Doravirine After Drug Intake Cessation up to 72 Hours Post-dose.
Description: Following cessation of daily dorivirine, plasm concentrations of drug to be taken were collected pre-dose and at 2,4,8, 12, 24, 30, 36, 48, 60 and 72h post-dose
Time Frame: 72 hours from treatment cessation; days 7-10 inclusive from enrolment
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Study Intervention
Number analyzed (Participants) | 14
ng*hr/mL
  t1/2 0-24h | 14.56 [13.19 to 16.59]
  t1/2 0-72h | 13.97 [12.77 to 15.68]

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: All adverse events to be recorded and reported during the study up to last visit.
Time Frame: From enrolment to last visit; last visit will be between days 20-23 from enrolment
Population: Safety and tolerability of study drug were investigated in population of participants for the study
Measure: Count of Participants; unit: Participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 14
Participants
  Hay Fever | 4
  Headache | 2
  No adverse events | 8

ADVERSE EVENTS:
Time Frame: Safety and tolerability of the studied drug was collected over a period of 23 days.
Description: All adverse events, however minor, were documented in the CRF whether or not the Investigator concludes the event to be related to drug treatment.
Arm/Group | Study Intervention
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Intervention (N=14)
Hay fever (Infections and infestations) | 4 (4)
Headaches (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03894124/Prot_SAP_000.pdf